CLINICAL TRIAL: NCT00059540
Title: The Maternal Lifestyle Study
Brief Title: The Maternal Lifestyle Study (MLS)
Acronym: MLS
Status: Completed | Type: Observational
Sponsor: NICHD Neonatal Research Network (Network)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH); Children's Bureau - Administration for Children and Families (Other); Substance Abuse and Mental Health Services Administration (SAMHSA) (U.S. Federal Agency); Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Sponsor
Other Study IDs: NICHD-NRN-0008; U10HD021397 (NIH); U10HD021415 (NIH); U10HD027904 (NIH); U10HD021385 (NIH); U10DA024117 (NIH); U10DA024118 (NIH); U10DA024119 (NIH); U10DA024128 (NIH)
Record Dates: First submitted 2003-04-28; First posted 2003-04-29 (Estimated); Last update posted 2016-09-21 (Estimated); Status verified 2016-09

CONDITIONS: Cocaine; Substance Abuse; Infant, Newborn; Pregnancy; Pregnant Women; Prenatal Care
Keywords: NICHD Neonatal Research Network; Maternal Lifestyle Study; Cocaine abuse; Cocaine dependence; Opiate abuse; Opiate dependence; Follow-up; Neurodevelopmental outcome; Substance-related disorders
MeSH Terms: conditions — Substance-Related Disorders; Cocaine-Related Disorders; Opioid-Related Disorders

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

SUMMARY:
This is a longitudinal, multi-site observational study of the long-term effects of a mother's use of cocaine and/or opiates during pregnancy on her infant. This observational study evaluates the medical, developmental, social, environmental, and neurobehavioral outcomes for 1,400 of the original cohort of children. A series of follow-up examinations of these children were conducted in 5 phases: 1-36 months, 3.5-7 years, and 8-11 years. Children are currently being examined at 13 years of age.

DETAILED DESCRIPTION:
Interest in and availability of cocaine, marijuana, and opiates have complicated long-term investigations into the effects of the widespread recreational use of easily accessible substances like alcohol and tobacco. It remains impossible to determine in single site, small number studies what effects may be related to the use of a specific drug. By accessing the large multi-site population of newborn infants and their mothers available in the NICHD Neonatal Research Network, this study is evaluating the short- and long-term effects of mothers' cocaine and/or opiate use during pregnancy on their term or preterm infants.

Maternal practices assessed in this study include the use and abuse of opiates, cocaine, alcohol, marijuana, and nicotine. This study will address acute perinatal events and long-term medical, developmental, social, environmental, and neurobehavioral outcomes of infants whose mothers engaged in these maternal practices. The study will determine whether specific acute and long-term effects can be attributed to the use and abuse of specific substances.

Over 2 years, approximately 20,000 infants were screened with a goal of enrolling 16,000 infants. It was estimated that approximately 20% of infants would have been exposed to cocaine or opiates. The determination of exposure was based on self-report by the mother or positive meconium assay.

The first phase of the study evaluated the acute effects of maternal practices on infants. This phase involved all mothers who agreed to respond to the initial questionnaire and who allowed the meconium drug screen to be performed on their infants. Acute outcomes are being compared between infants who were exposed to cocaine and opiates through their mothers' use (the exposed group) and infants who were not exposed (the nonexposed group). Acute outcomes include abruptio placenta, fetal growth retardation, non-life threatening congenital malformations, respiratory distress syndrome, chronic lung disease, periventricular-intraventricular hemorrhage, necrotizing enterocolitis, retinopathy of prematurity, and periventricular leukomalacia.

The second phase of the study compared 1,400 exposed and nonexposed infants with respect to long-term neurodevelopmental outcomes. These infants were among the 16,000 infants enrolled in Phase I. It was estimated that 70% of the screened population would consent to participate in Phase II of the study, and 50% of these participants would complete all visits over the initial 3-year study period (2,000 exposed infants enrolled into Phase II and 1,000 exposed infants would complete all follow-up visits). For each exposed infant, an infant of similar age, race, sex, and either alcohol history or maternal age was selected from the nonexposed, screened population. All infants had physical, neurological, gestational age, and growth assessments at birth. The exposed and nonexposed infants were examined at 1, 4, 7, 9, 12, 18, 24, and 36 months corrected age. Follow-up assessments include medical history, and developmental, behavioral, social, and environmental outcomes.

The third phase of the study compared children at ages 4 to 7. The fourth phase is now comparing outcomes in children ages 8 to 11 years old. Assessments include measures of cognition, school performance, antisocial behavior, onset of substance use, psychopathology, neuroendocrine function, and health disorders. Seventy-one percent of the original sample is still enrolled.

ELIGIBILITY:
Inclusion Criteria for Mothers:

* 18 years or older
* Live near a study site

Exclusion Criteria for Mothers:

* Identified psychosis or history of institutionalization for retardation or emotional problems
* Language barriers that prevented her from giving informed consent or understanding the study

Inclusion Criteria for Infants:

* Inborn infants
* Birthweight >501 grams (1.1 lbs)

Exclusion Criteria for Infants:

* One of a multiple gestation
* Gestational age >42 weeks
* Viability of the infant

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Mother and baby dyads delivered at the 4 participating centers.
Sampling Method: Non-Probability Sample
Enrollment: 11811 (Actual)
Dates: Start 1993-05; Primary Completion 1995-03 (Actual); Study Completion 2011-03 (Actual)

PRIMARY OUTCOMES:
Neurodevelopmental impairment | 1 month of age

CONTACTS AND LOCATIONS:
Overall Officials: Barry M. Lester, PhD, Principal Investigator — Brown University, Women & Infants Hospital of Rhode Island; Abhik Das, PhD, Principal Investigator — RTI International; Charles R. Bauer, MD, Principal Investigator — University of Miami; Henrietta S. Bada, MD, Principal Investigator — University of Tennessee; Seetha Shankaran, MD, Principal Investigator — Wayne State University
Locations (5):
- United States (5):
  - University of Miami, Miami, Florida
  - Wayne State University, Detroit, Michigan
  - RTI International, Durham, North Carolina
  - Brown University, Women & Infants Hospital of Rhode Island, Providence, Rhode Island
  - University of Tennessee, Memphis, Tennessee

REFERENCES:
- [Background] Lester BM, ElSohly M, Wright LL, Smeriglio VL, Verter J, Bauer CR, Shankaran S, Bada HS, Walls HH, Huestis MA, Finnegan LP, Maza PL. The Maternal Lifestyle Study: drug use by meconium toxicology and maternal self-report. Pediatrics. 2001 Feb;107(2):309-17. doi: 10.1542/peds.107.2.309. PMID 11158464
- [Background] Andreozzi L, Flanagan P, Seifer R, Brunner S, Lester B. Attachment classifications among 18-month-old children of adolescent mothers. Arch Pediatr Adolesc Med. 2002 Jan;156(1):20-6. doi: 10.1001/archpedi.156.1.20. PMID 11772186
- [Background] Bada HS, Bauer CR, Shankaran S, Lester B, Wright LL, Das A, Poole K, Smeriglio VL, Finnegan LP, Maza PL. Central and autonomic system signs with in utero drug exposure. Arch Dis Child Fetal Neonatal Ed. 2002 Sep;87(2):F106-12. doi: 10.1136/fn.87.2.f106. PMID 12193516
- [Background] Bada HS, Das A, Bauer CR, Shankaran S, Lester B, Wright LL, Verter J, Smeriglio VL, Finnegan LP, Maza PL. Gestational cocaine exposure and intrauterine growth: maternal lifestyle study. Obstet Gynecol. 2002 Nov;100(5 Pt 1):916-24. doi: 10.1016/s0029-7844(02)02199-3. PMID 12423853
- [Background] Bauer CR, Shankaran S, Bada HS, Lester B, Wright LL, Krause-Steinrauf H, Smeriglio VL, Finnegan LP, Maza PL, Verter J. The Maternal Lifestyle Study: drug exposure during pregnancy and short-term maternal outcomes. Am J Obstet Gynecol. 2002 Mar;186(3):487-95. doi: 10.1067/mob.2002.121073. PMID 11904612
- [Background] LaGasse LL, Messinger D, Lester BM, Seifer R, Tronick EZ, Bauer CR, Shankaran S, Bada HS, Wright LL, Smeriglio VL, Finnegan LP, Maza PL, Liu J. Prenatal drug exposure and maternal and infant feeding behaviour. Arch Dis Child Fetal Neonatal Ed. 2003 Sep;88(5):F391-9. doi: 10.1136/fn.88.5.f391. PMID 12937043
- [Background] Tronick EZ, Olson K, Rosenberg R, Bohne L, Lu J, Lester BM. Normative neurobehavioral performance of healthy infants on the Neonatal Intensive Care Unit Network Neurobehavioral Scale. Pediatrics. 2004 Mar;113(3 Pt 2):676-8. PMID 14993526
- [Background] Lester BM, Tronick EZ, LaGasse L, Seifer R, Bauer CR, Shankaran S, Bada HS, Wright LL, Smeriglio VL, Lu J. Summary statistics of neonatal intensive care unit network neurobehavioral scale scores from the maternal lifestyle study: a quasinormative sample. Pediatrics. 2004 Mar;113(3 Pt 2):668-75. PMID 14993525
- [Background] Lester BM, Tronick EZ, Brazelton TB. The Neonatal Intensive Care Unit Network Neurobehavioral Scale procedures. Pediatrics. 2004 Mar;113(3 Pt 2):641-67. PMID 14993524
- [Background] Lester BM, Tronick EZ. History and description of the Neonatal Intensive Care Unit Network Neurobehavioral Scale. Pediatrics. 2004 Mar;113(3 Pt 2):634-40. PMID 14993523
- [Background] Lester BM, Tronick EZ, LaGasse L, Seifer R, Bauer CR, Shankaran S, Bada HS, Wright LL, Smeriglio VL, Lu J, Finnegan LP, Maza PL. The maternal lifestyle study: effects of substance exposure during pregnancy on neurodevelopmental outcome in 1-month-old infants. Pediatrics. 2002 Dec;110(6):1182-92. doi: 10.1542/peds.110.6.1182. PMID 12456917
- [Background] Lester BM, Lagasse L, Seifer R, Tronick EZ, Bauer CR, Shankaran S, Bada HS, Wright LL, Smeriglio VL, Liu J, Finnegan LP, Maza PL. The Maternal Lifestyle Study (MLS): effects of prenatal cocaine and/or opiate exposure on auditory brain response at one month. J Pediatr. 2003 Mar;142(3):279-85. doi: 10.1067/mpd.2003.112. PMID 12640376
- [Background] Messinger DS, Bauer CR, Das A, Seifer R, Lester BM, Lagasse LL, Wright LL, Shankaran S, Bada HS, Smeriglio VL, Langer JC, Beeghly M, Poole WK. The maternal lifestyle study: cognitive, motor, and behavioral outcomes of cocaine-exposed and opiate-exposed infants through three years of age. Pediatrics. 2004 Jun;113(6):1677-85. doi: 10.1542/peds.113.6.1677. PMID 15173491
- [Background] Seifer R, LaGasse LL, Lester B, Bauer CR, Shankaran S, Bada HS, Wright LL, Smeriglio VL, Liu J. Attachment status in children prenatally exposed to cocaine and other substances. Child Dev. 2004 May-Jun;75(3):850-68. doi: 10.1111/j.1467-8624.2004.00710.x. PMID 15144490
- [Background] Shankaran S, Das A, Bauer CR, Bada HS, Lester B, Wright LL, Smeriglio V. Association between patterns of maternal substance use and infant birth weight, length, and head circumference. Pediatrics. 2004 Aug;114(2):e226-34. doi: 10.1542/peds.114.2.e226. PMID 15286261
- [Background] Shankaran S, Bauer CR, Bada HS, Lester B, Wright LL, Das A. Health-care utilization among mothers and infants following cocaine exposure. J Perinatol. 2003 Jul-Aug;23(5):361-7. doi: 10.1038/sj.jp.7210946. PMID 12847529
- [Background] Das A, Poole WK, Bada HS. A repeated measures approach for simultaneous modeling of multiple neurobehavioral outcomes in newborns exposed to cocaine in utero. Am J Epidemiol. 2004 May 1;159(9):891-9. doi: 10.1093/aje/kwh114. PMID 15105182
- [Background] Boukydis CF, Bigsby R, Lester BM. Clinical use of the Neonatal Intensive Care Unit Network Neurobehavioral Scale. Pediatrics. 2004 Mar;113(3 Pt 2):679-89. PMID 14993527
- [Result] Bada HS, Das A, Bauer CR, Shankaran S, Lester B, LaGasse L, Hammond J, Wright LL, Higgins R. Impact of prenatal cocaine exposure on child behavior problems through school age. Pediatrics. 2007 Feb;119(2):e348-59. doi: 10.1542/peds.2006-1404. PMID 17272597
- [Result] Bada HS, Bann CM, Bauer CR, Shankaran S, Lester B, LaGasse L, Hammond J, Whitaker T, Das A, Tan S, Higgins R. Preadolescent behavior problems after prenatal cocaine exposure: Relationship between teacher and caretaker ratings (Maternal Lifestyle Study). Neurotoxicol Teratol. 2011 Jan-Feb;33(1):78-87. doi: 10.1016/j.ntt.2010.06.005. Epub 2010 Jun 30. PMID 20600844
- [Result] Bada HS, Bauer CR, Shankaran S, Lester B, Wright LL, Verter J, Smeriglio VL, Finnegan LP, Maza PL. Central and autonomic nervous systems' signs associated with in utero exposure to cocaine/opiates. Ann N Y Acad Sci. 1998 Jun 21;846:431-4. PMID 9668443
- [Result] Bada HS, Das A, Bauer CR, Shankaran S, Lester BM, Gard CC, Wright LL, Lagasse L, Higgins R. Low birth weight and preterm births: etiologic fraction attributable to prenatal drug exposure. J Perinatol. 2005 Oct;25(10):631-7. doi: 10.1038/sj.jp.7211378. PMID 16107872
- [Result] Bada HS, Langer J, Twomey J, Bursi C, Lagasse L, Bauer CR, Shankaran S, Lester BM, Higgins R, Maza PL. Importance of stability of early living arrangements on behavior outcomes of children with and without prenatal drug exposure. J Dev Behav Pediatr. 2008 Jun;29(3):173-82. doi: 10.1097/DBP.0b013e3181644a79. PMID 18349707
- [Result] Bagner DM, Sheinkopf SJ, Miller-Loncar C, LaGasse LL, Lester BM, Liu J, Bauer CR, Shankaran S, Bada H, Das A. The effect of parenting stress on child behavior problems in high-risk children with prenatal drug exposure. Child Psychiatry Hum Dev. 2009 Mar;40(1):73-84. doi: 10.1007/s10578-008-0109-6. Epub 2008 Jul 15. PMID 18626768
- [Result] Bauer CR, Langer JC, Shankaran S, Bada HS, Lester B, Wright LL, Krause-Steinrauf H, Smeriglio VL, Finnegan LP, Maza PL, Verter J. Acute neonatal effects of cocaine exposure during pregnancy. Arch Pediatr Adolesc Med. 2005 Sep;159(9):824-34. doi: 10.1001/archpedi.159.9.824. PMID 16143741
- [Result] ElSohly MA, Stanford DF, Murphy TP, Lester BM, Wright LL, Smeriglio VL, Verter J, Bauer CR, Shankaran S, Bada HS, Walls HC. Immunoassay and GC-MS procedures for the analysis of drugs of abuse in meconium. J Anal Toxicol. 1999 Oct;23(6):436-45. doi: 10.1093/jat/23.6.436. PMID 10517548
- [Result] Gaskins RB, LaGasse LL, Liu J, Shankaran S, Lester BM, Bada HS, Bauer CR, Das A, Higgins RD, Roberts M. Small for gestational age and higher birth weight predict childhood obesity in preterm infants. Am J Perinatol. 2010 Oct;27(9):721-30. doi: 10.1055/s-0030-1253555. Epub 2010 Apr 20. PMID 20408111
- [Result] Gauthier SM, Bauer CR, Messinger DS, Closius JM. The Bayley Scales of Infant Development. II: Where to start? J Dev Behav Pediatr. 1999 Apr;20(2):75-9. doi: 10.1097/00004703-199904000-00001. PMID 10219684
- [Result] LaGasse LL, Van Vorst RF, Brunner SM, Lester BM. Effects of in utero exposure to cocaine and/or opiates on infants' reaching behavior. Ann N Y Acad Sci. 1998 Jun 21;846:405-7. No abstract available. PMID 9668436
- [Result] Sheinkopf SJ, Lagasse LL, Lester BM, Liu J, Seifer R, Bauer CR, Shankaran S, Bada H, Higgins R, DAS A. Prenatal cocaine exposure: cardiorespiratory function and resilience. Ann N Y Acad Sci. 2006 Dec;1094:354-8. doi: 10.1196/annals.1376.049. PMID 17347376
- [Result] Lester BM. The Maternal Lifestyles Study. Ann N Y Acad Sci. 1998 Jun 21;846:296-305. No abstract available. PMID 9668416
- [Result] Lester BM, Bagner DM, Liu J, LaGasse LL, Seifer R, Bauer CR, Shankaran S, Bada H, Higgins RD, Das A. Infant neurobehavioral dysregulation: behavior problems in children with prenatal substance exposure. Pediatrics. 2009 Nov;124(5):1355-62. doi: 10.1542/peds.2008-2898. Epub 2009 Oct 12. PMID 19822596
- [Result] Lester BM, Lagasse LL, Shankaran S, Bada HS, Bauer CR, Lin R, Das A, Higgins R. Prenatal cocaine exposure related to cortisol stress reactivity in 11-year-old children. J Pediatr. 2010 Aug;157(2):288-295.e1. doi: 10.1016/j.jpeds.2010.02.039. Epub 2010 Apr 18. PMID 20400094
- [Result] Levine TP, Liu J, Das A, Lester B, Lagasse L, Shankaran S, Bada HS, Bauer CR, Higgins R. Effects of prenatal cocaine exposure on special education in school-aged children. Pediatrics. 2008 Jul;122(1):e83-91. doi: 10.1542/peds.2007-2826. Epub 2008 Jun 9. PMID 18541617
- [Result] Liu J, Bann C, Lester B, Tronick E, Das A, Lagasse L, Bauer C, Shankaran S, Bada H. Neonatal neurobehavior predicts medical and behavioral outcome. Pediatrics. 2010 Jan;125(1):e90-8. doi: 10.1542/peds.2009-0204. Epub 2009 Dec 7. PMID 19969621
- [Result] Maza PL, Wright LL, Bauer CR, Shankaran S, Bada HS, Lester B, Krause-Steinrauf H, Smeriglio VL, Bowler A, Katsikiotis V. Maternal Lifestyles Study (MLS). Caretaking environment and stability of substance-exposed infants at one month corrected age. Ann N Y Acad Sci. 1998 Jun 21;846:358-61. No abstract available. PMID 9668424
- [Result] Miller-Loncar C, Lester BM, Seifer R, Lagasse LL, Bauer CR, Shankaran S, Bada HS, Wright LL, Smeriglio VL, Bigsby R, Liu J. Predictors of motor development in children prenatally exposed to cocaine. Neurotoxicol Teratol. 2005 Mar-Apr;27(2):213-20. doi: 10.1016/j.ntt.2004.10.007. Epub 2004 Nov 25. PMID 15734272
- [Result] Salisbury AL, Lester BM, Seifer R, Lagasse L, Bauer CR, Shankaran S, Bada H, Wright L, Liu J, Poole K. Prenatal cocaine use and maternal depression: effects on infant neurobehavior. Neurotoxicol Teratol. 2007 May-Jun;29(3):331-40. doi: 10.1016/j.ntt.2006.12.001. Epub 2006 Dec 14. PMID 17258430
- [Result] Shankaran S, Das A, Bauer CR, Bada H, Lester B, Wright L, Higgins R, Poole K. Fetal origin of childhood disease: intrauterine growth restriction in term infants and risk for hypertension at 6 years of age. Arch Pediatr Adolesc Med. 2006 Sep;160(9):977-81. doi: 10.1001/archpedi.160.9.977. PMID 16953023
- [Result] Shankaran S, Lester BM, Das A, Bauer CR, Bada HS, Lagasse L, Higgins R. Impact of maternal substance use during pregnancy on childhood outcome. Semin Fetal Neonatal Med. 2007 Apr;12(2):143-50. doi: 10.1016/j.siny.2007.01.002. Epub 2007 Feb 20. PMID 17317350
- [Result] Sheinkopf SJ, Lagasse LL, Lester BM, Liu J, Seifer R, Bauer CR, Shankaran S, Bada H, Das A. Vagal tone as a resilience factor in children with prenatal cocaine exposure. Dev Psychopathol. 2007 Summer;19(3):649-73. doi: 10.1017/S0954579407000338. PMID 17705897
- [Result] Sheinkopf SJ, Lester BM, LaGasse LL, Seifer R, Bauer CR, Shankaran S, Bada HS, Poole WK, Wright LL. Interactions between maternal characteristics and neonatal behavior in the prediction of parenting stress and perception of infant temperament. J Pediatr Psychol. 2006 Jan-Feb;31(1):27-40. doi: 10.1093/jpepsy/jsj026. Epub 2005 Apr 12. PMID 15827350
- [Result] Sheinkopf SJ, Lester BM, Sanes JN, Eliassen JC, Hutchison ER, Seifer R, Lagasse LL, Durston S, Casey BJ. Functional MRI and response inhibition in children exposed to cocaine in utero. Preliminary findings. Dev Neurosci. 2009;31(1-2):159-66. doi: 10.1159/000207503. Epub 2009 Apr 17. PMID 19372696
- [Result] Stephens BE, Liu J, Lester B, Lagasse L, Shankaran S, Bada H, Bauer C, Das A, Higgins R. Neurobehavioral assessment predicts motor outcome in preterm infants. J Pediatr. 2010 Mar;156(3):366-71. doi: 10.1016/j.jpeds.2009.09.042. Epub 2009 Nov 1. PMID 19880137
- [Result] Stone KC, High PC, Miller-Loncar CL, Lagasse LL, Lester BM. Longitudinal study of maternal report of sleep problems in children with prenatal exposure to cocaine and other drugs. Behav Sleep Med. 2009;7(4):196-207. doi: 10.1080/15402000903190108. PMID 19787489
- [Result] Stone KC, LaGasse LL, Lester BM, Shankaran S, Bada HS, Bauer CR, Hammond JA. Sleep problems in children with prenatal substance exposure: the Maternal Lifestyle study. Arch Pediatr Adolesc Med. 2010 May;164(5):452-6. doi: 10.1001/archpediatrics.2010.52. PMID 20439796